CLINICAL TRIAL: NCT07110558
Title: A Single-arm, Phase II Trial of Radiotherapy Without Prophylactic Neck Irradiation in Combination With Neoadjuvant and Adjuvant Anti-PD-1 Antibody Toripalimab for Nasopharyngeal Carcinoma
Brief Title: Radiotherapy Omitting Prophylactic Neck Irradiation With Neoadjuvant and Adjuvant Toripalimab in Nasopharyngeal Carcinoma
Acronym: PUPA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-068
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; radiotherapy; immunotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Toripalimab group (Experimental): NPC Patients without cervical lymph node metastasis (N0 or N1 restricted to retropharyngeal lymph nodes) received two cycles of toripalimab, followed by cisplatin concurrent chemoradiotherapy without prophylactic neck irradiation, and adjuvant toripalimab up to 8 cycles.
  Interventions: Radiation: Without prophylactic neck irradiation; Drug: PD-1 antibody (Toripalimab); Drug: Cisplatin

INTERVENTIONS:
Radiation: Without prophylactic neck irradiation — Intensity-modulated radiotherapy restricted to the primary tumor, omitting prophylactic neck irradiation.
Drug: PD-1 antibody (Toripalimab) — Toripalimab 240mg every 2 weeks with a total of 2 cycles as neoadjuvant anti-PD-1 immunotherapy; Toripalimab 240mg every 3 weeks with a total of 8 cycles as adjuvant anti-PD-1 immunotherapy after CCRT
Drug: Cisplatin — Cisplatin 100mg/m2(every three weeks), Day 1, Day 22, Day 43 of intensity modulated radiotherapy

SUMMARY:
This single-arm, phase 2 trial evaluates the efficacy and safety of de-escalated radiotherapy (restricted to the primary tumor, omitting prophylactic neck irradiation) combined with neoadjuvant and adjuvant toripalimab immunotherapy, and concurrent chemotherapy in patients with nasopharyngeal carcinoma staged N0 or N1, where nodal involvement is strictly confined to the retropharyngeal lymph nodes.

DETAILED DESCRIPTION:
The goals of this clinical trial includes: ① To assess the regional relapse-free survival (RRFS) and safety after radiotherapy without prophylactic neck irradiation in combination with neoadjuvant and adjuvant PD-1 antibody toripalimab and cisplatin concurrent chemotherapy for N0-1 (restricted to retropharyngeal lymph nodes) patients with nasopharyngeal carcinoma; ② To evaluate the impact of radiotherapy without prophylactic neck irradiation on 2-year overall survival (OS), 2-year progress-free survival (PFS), 2-year distant metastasis-free survival (DMFS), and 2-year locoregional relapse-free survival (LRRFS) for N0-1 ( limited to retropharyngeal lymph nodes) patients with nasopharyngeal carcinoma; ③ To explore the impact of radiotherapy without prophylactic neck irradiation on toxicities and quality of life; ④ To explore the relationship between clinical factors and the impact of neoadjuvant and adjuvant PD-1 antibody, radiotherapy without prophylactic neck irradiation on the survival of patients; ⑤ To explore the biomarkers of sensitivity to immunotherapy, chemotherapy and radiotherapy for patients with nasopharyngeal carcinoma and the underlying mechanism.

For these purposes, we plan to prospectively enroll T2N0-1 and primary gross tumor volume (GTV) greater than 30.0 cm3 or T3-4N0-1 stage NPC patients, whose N1 restricted to retropharyngeal lymph nodes from one center in China. The patients will receive 2 cycles of neoadjuvant PD-1 antibody (toripalimab monotherapy, 240 mg, every two weeks, intravenous infusion) followed by concurrent cisplatin (100 mg/m2 intravenously) on days 1, 22, and 43 during intensity-modulated radiotherapy (IMRT), and adjuvant toripalimab (240 mg intravenously) once every 3 weeks for up to eight cycles. All participants will be treated with IMRT restricted to primary tumor without prophylactic neck irradiation. The clinical outcomes, safety, complications, and quality of life will be explored in the RT without prophylactic neck irradiation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 Years to 70 Years;
2. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
3. Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1
4. TNM stage based on AJCC 9th edition with N0-1 (retroperitoneal lymph nodes only), and either one following criteria:

   1. T2 and primary gross tumor volume (GTV) greater than 30.0 cm3;
   2. T3-4;
5. Patients' lymph node without adverse features (no central necrosis, no muscle/skin invasion, no lymph node fusion).
6. Male and no pregnant female
7. Normal bone marrow function: white blood cell count > 4×10^9/L, hemoglobin > 90g/L, platelet count > 100×10^9/L;
8. Normal liver function: total bilirubin (TBIL) < upper limit of normal (ULN), alanine transaminase (ALT) and aspartate transaminase (AST) < 1.5 × ULN;
9. Normal kidney function: creatinine clearance rate ≥ 60 ml/min;
10. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;

Exclusion Criteria:

1. Patients have evidence of relapse or distant metastasis
2. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
3. Patients with positive cervical lymph nodes
4. Patients who have been treated with inhibitors of immune regulation (CTLA-4, PD-1, PD-L1, etc.).
5. Receiving radiotherapy or chemotherapy previously
6. Patients with active immunodeficiency disease and history of immunodeficiency disease
7. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS)
8. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible.
9. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment, history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved.
10. HBV DNA >2000 cps/ml (or HBV DNA > 2000 IU/ml); or HCV RNA >1000 cps/ml; Hepatitis B surface antigen (HBsAg) positive and HCV antibody positive.
11. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
12. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
13. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2), 2) unstable angina, 3) myocardial infarction in past 1 year, 4) supraventricular or ventricular arrhythmia requiring treatment or intervention.
14. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
15. Severe, uncontrolled medical conditions and infections.
16. At the same time using other test drugs or in other clinical trials.
17. Refusal or inability to sign informed consent to participate in the trial.
18. Other treatment contraindications.
19. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2029-08-14 (Estimated); Study Completion 2032-08-14 (Estimated)

PRIMARY OUTCOMES:
Regional relapse-free survival (RRFS) | 2 years
  Defined as the time from registration to documented nodal relapse or non-cancer-specific death.

SECONDARY OUTCOMES:
Progress-free survival (PFS) | 2 years
  Defined as the time from registration to documented disease progression or non-cancer-specific death.
Overall Survival (OS) | 2 years
  Defined as the time from registration to death from any cause.
Locoregional Relapse-Free Survival (LRRFS) | 2 years
  Defined as the time from registration to documented locoregional recurrence or non-cancer-specific death.
Distant Metastasis-Free Survival (DMFS) | 2 years
  Defined from registration to documented distant metastasis or noncancer-specific death.
Objective Response Rate （ORR） | After the completion of the neoadjuvant PD-1 antibody and chemoradiotherapy treatment
  An objective response is defined as either a confirmed CR or a PR, as determined by the investigator using RECIST v1.1Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI).
Incidence rate of acute and late adverse events (AEs) | 2 years
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. Acute AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0 (CTCAE 5.0). Late radiation toxicities were assessed using the Radiation Therapy Oncology Group (RTOG) and European Organisation for Research and Treatment of Cancer (EORTC).
Change of QoL (quality of life) | 1 year
  QoL scores were assessed by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) and Quality-of-Life Head and Neck 35 items (QLQ-H&N35) before neoadjuvant PD-1 antibody, before radiotherapy, at the end of radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, MD,PhD, Principal Investigator — Sun Yat-sen Universitty Cancer Center
Locations (1):
- Sun Yat-sen Universitty Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted to the Research Data Deposit (RDD) public platform (http://www.researchdata.org.cn) and available from the principal investigators upon reasonable request.

REFERENCES:
- [Background] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Background] Patel SP, Othus M, Chen Y, Wright GP Jr, Yost KJ, Hyngstrom JR, Hu-Lieskovan S, Lao CD, Fecher LA, Truong TG, Eisenstein JL, Chandra S, Sosman JA, Kendra KL, Wu RC, Devoe CE, Deutsch GB, Hegde A, Khalil M, Mangla A, Reese AM, Ross MI, Poklepovic AS, Phan GQ, Onitilo AA, Yasar DG, Powers BC, Doolittle GC, In GK, Kokot N, Gibney GT, Atkins MB, Shaheen M, Warneke JA, Ikeguchi A, Najera JE, Chmielowski B, Crompton JG, Floyd JD, Hsueh E, Margolin KA, Chow WA, Grossmann KF, Dietrich E, Prieto VG, Lowe MC, Buchbinder EI, Kirkwood JM, Korde L, Moon J, Sharon E, Sondak VK, Ribas A. Neoadjuvant-Adjuvant or Adjuvant-Only Pembrolizumab in Advanced Melanoma. N Engl J Med. 2023 Mar 2;388(9):813-823. doi: 10.1056/NEJMoa2211437. PMID 36856617
- [Background] Tang LL, Huang CL, Zhang N, Jiang W, Wu YS, Huang SH, Mao YP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Sun Y, Xie FY, Chen L, Zhou GQ, Ma J. Elective upper-neck versus whole-neck irradiation of the uninvolved neck in patients with nasopharyngeal carcinoma: an open-label, non-inferiority, multicentre, randomised phase 3 trial. Lancet Oncol. 2022 Apr;23(4):479-490. doi: 10.1016/S1470-2045(22)00058-4. Epub 2022 Feb 28. PMID 35240053
- [Background] Mai HQ, Chen QY, Chen D, Hu C, Yang K, Wen J, Li J, Shi Y, Jin F, Xu R, Pan J, Qu S, Li P, Hu C, Liu YC, Jiang Y, He X, Wang HM, Lim WT, Liao W, He X, Chen X, Wang S, Yuan X, Li Q, Lin X, Jing S, Chen Y, Lu Y, Hsieh CY, Yang MH, Yen CJ, Samol J, Luo X, Wang X, Tang X, Feng H, Yao S, Keegan P, Xu RH. Toripalimab Plus Chemotherapy for Recurrent or Metastatic Nasopharyngeal Carcinoma: The JUPITER-02 Randomized Clinical Trial. JAMA. 2023 Nov 28;330(20):1961-1970. doi: 10.1001/jama.2023.20181. PMID 38015220
- [Background] Liu SL, Li XY, Yang JH, Wen DX, Guo SS, Liu LT, Li YF, Luo MJ, Xie SY, Liang YJ, Sun XS, Yang ZC, Lv XF, Luo DH, Li JB, Liu Q, Wang P, Guo L, Mo HY, Sun R, Yang Q, Lan KQ, Jia GD, Li R, Zhao C, Xu RH, Chen QY, Tang LQ, Mai HQ. Neoadjuvant and adjuvant toripalimab for locoregionally advanced nasopharyngeal carcinoma: a randomised, single-centre, double-blind, placebo-controlled, phase 2 trial. Lancet Oncol. 2024 Dec;25(12):1563-1575. doi: 10.1016/S1470-2045(24)00504-7. Epub 2024 Nov 7. PMID 39522541